CLINICAL TRIAL: NCT02400567
Title: Open-label, Randomized, Multicenter, International, Parallel Exploratory Phase II Study, Comparing 3 FEC-3 Docetaxel Chemotherapy to Letrozole + Palbociclib Combination as Neoadjuvant Treatment of Stage II-IIIA PAM 50 ROR-defined Low or Intermediate Risk Luminal Breast Cancer, in Postmenopausal Women
Brief Title: Efficacy of Letrozole + Palbociclib Combination as Neoadjuvant Treatment of Stage II-IIIA PAM 50 ROR-defined Low or Intermediate Risk Luminal Breast Cancer, in Postmenopausal Women
Acronym: NeoPAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Pfizer (Industry); NanoString Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeoPal - UC-0140/1404; 2014-002560-33 (EudraCT Number); CARMINA04 (Other: UNICANCER); NEOPAL (Other: UNICANCER)
Record Dates: First submitted 2014-08-05; First posted 2015-03-27 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Neoadjuvant Operable Breast Cancer
Keywords: Luminal; Post menopausal; Breast conservation; Neoadjuvant
MeSH Terms: interventions — Fluorouracil; Epirubicin; Cyclophosphamide; Letrozole; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Active Comparator): 3 cycles of FEC 100 followed by 3 cycles of Docetaxel Drugs: Fluorouracile, Epirubicine, Cyclophosphamide, Docetaxel
  Interventions: Drug: Fluorouracile; Drug: Epirubicin; Drug: Cyclophosphamide
- Letrozole Palbociclib (Experimental): Drugs: letrozole + palbociclib combination
  Interventions: Drug: Letrozole; Drug: Palbociclib

INTERVENTIONS:
Drug: Fluorouracile
  Arms: Chemotherapy
Drug: Epirubicin
  Arms: Chemotherapy
Drug: Cyclophosphamide
  Arms: Chemotherapy
Drug: Letrozole
  Arms: Letrozole Palbociclib
Drug: Palbociclib
  Arms: Letrozole Palbociclib

SUMMARY:
The investigators propose in the present study an innovative approach, combining the most recent therapeutic opportunities in high risk ER+ breast cancer with the most recent and innovative diagnostic approaches such as the PAM50 signature and the RCB tumor response evaluation method. In line with the most recent recommendations on targeted anticancer therapies, the investigators have designed a parallel phase II randomized trial with early stopping rules 26, which will able in the meantime to build a unique prospective collection of tumor tissue, pre- and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years, Post-menopausal women
2. Newly diagnosed and operable unilateral invasive breast cancer, not candidate or uncertain for breast conservation - Note: Multicentric/multifocal tumors are allowed provided a maximum of 3 lesions are present, and all share the same characteristics: ER Allred 4, Her2- (PAM50 will be performed in the largest lesion)
3. Stage II-IIIA
4. Assessment of nodal status available (Ultrasound guided FNA or biopsy if necessary)
5. Non metastatic, M0
6. ER-positive by IHC (Allred Score≥4)
7. HER2-negative by IHC (score 0 or 1+) and/or Fish/Cish
8. Either Luminal A AND proven nodal involvement (cytology or histology), or Luminal B through PAM50 ROR (Prosigna™) centralized evaluation
9. ECOG 0-1
10. No prior systemic therapy for the present tumor
11. Adequate renal, hepatic, and hematopoietic functions as defined by the following criteria:

    * Absolute Neutrophil Count (ANC) ≥1,500/mm3 or ≥1.5 x 109/L
    * Platelets ≥100,000/mm3 or ≥100 x 109/L
    * Hemoglobin ≥9 g/dL
    * Serum Aspartate Transaminase (AST) and serum Alanine Aminotransferase Transaminase (ALT) ≤2.5 x upper limit of normal (ULN)
    * Alkaline phosphatase ≤2.5 x ULN
    * Total serum bilirubin ≤1 x ULN
    * Serum creatinine ≤1.5 x ULN or estimated creatinine clearance ≥ 60 mL/min as calculated using the method standard for the institution
12. Adequate cardiac functions, including:

    * 12 Lead electrocardiogram (ECG) with normal tracing or non clinically significant changes that do not require medical intervention.
    * QTc interval ≤480 msec
    * No history of Torsades de Pointes or other symptomatic QTc abnormality.
13. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures
14. Signed informed consent and health insurance coverage

Exclusion Criteria:

1. Non operable, bilateral, T4 or metastatic breast cancer
2. Limited T2 breast cancer immediately accessible to conservative surgery
3. Previous homolateral breast cancer (including in situ carcinoma), and/or contralateral breast cancer except if treated by surgery +/- radiation therapy alone without any systemic treatment
4. Previous hormone replacement therapy (HRT) stopped less than 2 weeks before beginning of treatment
5. Previous use of SERMs such as raloxifene
6. Any surgery (not including minor procedures such as lymph node biopsy, primary tumor core biopsy, fine needle aspiration) within 4 weeks of start of study treatment; or not fully recovered from any side effects of previous procedures.
7. Diagnosis of any previous malignancy within the last 5 years, except for adequately treated basal cell carcinoma, or squamous cell skin carcinoma, or in situ cervical carcinoma
8. History of any previous anti-cancer chemotherapy and any previous treatment using AI
9. Concurrent administration of herbal preparations as complementary medicine.
10. Any clinically significant gastrointestinal abnormalities, which may impair intake, transit or absorption of the study drugs, such as the inability to take oral medication in tablet form and malabsorption syndrome
11. Patient with any psychological, familial, social or geographical condition which could potentially hamper compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the number of patients with a Residual Cancer Burden (RCB) 0-I index as a measure of efficacy | 21 weeks
  Residual cancer burden (RCB) is estimated from routine pathologic sections of the primary breast tumor site and the regional lymph nodes after the completion of neoadjuvant therapy. 6 variables are included in a calculation formula.

SECONDARY OUTCOMES:
Evaluation of the clinical response in each treatment arm as defined by clinical and ultrasound examination. | 21 weeks
Determination of the number and type of Adverse Events as a Measure of Safety and Tolerability | 21 weeks
  The toxicity will be evaluated according to the scale CTC-AE version 4.0
Correlation of the PAM50 risk of recurrence (ROR) score to its ability to predict RCB as defined in outcome 1 | 21 weeks
Calculation of the rates of breast conservation therapy in the two arms with regard to the initially planned surgery. | 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cottu, MD, Principal Investigator — Institut Curie Paris; Suzette Delaloge, MD, Principal Investigator — Gustave roussy, Villejuif
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Result] Cottu P, D'Hondt V, Dureau S, Lerebours F, Desmoulins I, Heudel PE, Duhoux FP, Levy C, Mouret-Reynier MA, Dalenc F, Frenel JS, Jouannaud C, Venat-Bouvet L, Nguyen S, Ferrero JM, Canon JL, Grenier J, Callens C, Gentien D, Lemonnier J, Vincent-Salomon A, Delaloge S. Letrozole and palbociclib versus chemotherapy as neoadjuvant therapy of high-risk luminal breast cancer. Ann Oncol. 2018 Dec 1;29(12):2334-2340. doi: 10.1093/annonc/mdy448. PMID 30307466
- See also: Ann Oncol . 2018 Dec 1;29(12):2334-2340. doi: 10.1093/annonc/mdy448 — https://pubmed.ncbi.nlm.nih.gov/30307466/